CLINICAL TRIAL: NCT04782804
Title: Adjuvant PD-1 Antibody（Tislelizumab） in Combination With Capecitabine for Patients With Cholangiocarcinoma at High-Risk of Postoperative Recurrence
Brief Title: Adjuvant PD-1 Antibody in Combination With Capecitabine for Patients With ICC at High-Risk of Postoperative Recurrence
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, Director of the general surgery department, Huashan hospital, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUASHAN006
Record Dates: First submitted 2021-03-03; First posted 2021-03-04 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Cholangiocarcinoma, Intrahepatic
Keywords: Cholangiocarcinoma; PD1; adjuvant therapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Capecitabine; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine (Active Comparator): Capecitabine as Adjuvant Therapy Oral capecitabine (1250 mg/m²) was given post operatively twice a day on days 1 to 14 of a 3-weekly cycle for 24 weeks (eight cycles), and observation commenced within 16 weeks of surgery.
  Interventions: Drug: Capecitabine
- Capecitabine+PD-1 Antibody（Tislelizumab） (Experimental): Capecitabine+PD-1 Antibody（Tislelizumab）as Adjuvant Therapy Oral capecitabine (1250 mg/m²) was given post operatively twice a day on days 1 to 14 of a 3-weekly cycle for 24 weeks (eight cycles), and observation commenced within 16 weeks of surgery. PD-1 Antibody（Tislelizumab, 200mg） was given q3w iv.
  Interventions: Drug: Capecitabine; Drug: PD-1 Antibody（Tislelizumab）

INTERVENTIONS:
Drug: Capecitabine — Capecitabine+PD-1 Antibody（Tislelizumab）as Adjuvant Therapy Oral capecitabine (1250 mg/m²) was given post operatively twice a day on days 1 to 14 of a 3-weekly cycle for 24 weeks (eight cycles), and observation commenced within 16 weeks of surgery.
  Other Names: XELODA
Drug: PD-1 Antibody（Tislelizumab） — PD-1 Antibody（Tislelizumab, 200mg） was given q3w iv.
  Other Names: Tislelizumab
  Arms: Capecitabine+PD-1 Antibody（Tislelizumab）

SUMMARY:
The purpose of the study is to observe the effect of PD-1 Antibody（Tislelizumab） Combined With Capecitabine as Adjuvant Therapy to Prevent the Recurrence in High-risk Patients With Cholangiocarcinoma After Curative Resection.

DETAILED DESCRIPTION:
Cholangiocarcinoma has a low incidence, accounting for only 3% of gastrointestinal malignancies worldwide, but with an increasing trend in recent years.Cholangiocarcinoma is extremely malignant, and the 5-year survival rate for patients who cannot undergo curative resection at advanced stages is less than 10%. Surgical resection represents the only curative opportunity for biliary tract cancer, but only 1 5% - 20% of patients can undergo surgical resection; however, even patients who undergo curative surgical resection have a high rate of postoperative metastasis recurrence, and effective treatment strategies are lacking after metastasis recurrence.The median postoperative survival time is only 18-30 months and the 5-year survival rate is also only 20-35%.Among them, patients with high-risk postoperative recurrence who are resected but have positive lymph nodes or margins have further reduced survival, and no targeted effective postoperative adjuvant therapy is available, becoming another important reason that hampers the long-term survival of surgical patients.

For unresectable or advanced cholangiocarcinoma, GEMOX, a two drug combination regimen of gemcitabine plus cisplatin, can be used as a first-line chemotherapy regimen, but the first-line regimen of postoperative adjuvant chemotherapy is currently not uniformly recommended.Previous adjuvant chemotherapy for cholangiocarcinoma was mostly based on clinical experience from different medical centers and borrowed in view of gemcitabine - and platinum based advanced regimens, but the conclusions based on retrospective studies varied greatly among different centers and the recommendation was limited.Whereas there are fewer prospective studies aiming to target postoperative adjuvant chemotherapy for cholangiocarcinoma.The 2017 Prodige prospective randomized controlled study evaluated the efficacy of GEMOX in advanced cholangiocarcinoma in 196 patients treated with postoperative adjuvant chemotherapy and showed that although there was a trend toward benefit in RFs, it was not statistically significant overall and does not support the use of the GEMOX regimen in advanced cholangiocarcinoma in the postoperative adjuvant setting.While another 2018 bcat prospective study negated the clinical benefit of gemcitabine monotherapy in postoperative adjuvant chemotherapy for cholangiocarcinoma.In contrast, the 2017 Bilcap study was the only one to yield positive results in postoperative adjuvant chemotherapy for cholangiocarcinoma.The study compared the clinical value of capecitabine with clinical observation in postoperative adjuvant chemotherapy for cholangiocarcinoma, the primary endpoint was OS, the secondary endpoints included OS, recurrence free survival (RFs), etc. adjuvant capecitabine can extend the OS of postoperative cholangiocarcinoma from 36 to 51 months, and in terms of safety, the differences in toxicity between the capecitabine combination control groups were not significant and most of themNumber patients could tolerate.Therefore, the ASCO guidelines also recommend adjuvant chemotherapy with capecitabine in patients with cholangiocarcinoma after surgery and recommend it as a control for subsequent clinical studies in cholangiocarcinoma.However, whether capecitabine monotherapy can play a role in preventing recurrence in patients with high-risk disease who have undergone surgery with positive lymph nodes or resection margins remains to be confirmed by further studies.

Cholangiocarcinoma is accompanied by a dysregulation and remodelling of the local immune microenvironment, and therefore the catalysed tumour immunotherapy has been a long-standing hotspot in the field of cancer therapy, in which T-cell-based tumour immunotherapy is in its core position. 1 cancer immunotherapy is fully used and mobilising killer T cells from the tumour bearing patient. 2Cells, to carry out the killing effect on the tumor, it may be the most effective and the safest way to treat the tumor.At the same time, tumor escape is a formidable obstacle facing tumor immunotherapy, in which tumor cells exploit their own suppressive effects on the immune system to promote deranged tumor growth.There is an extremely complex relationship between the immune escape mechanism of tumors and the host immune response to tumors.Tumor immunotherapy tumor specific killer T cells in the early stage are biologically active, but lose the function of killing as the tumor grows later.So tumor immunotherapy is to maximize the patient's own immune system reaction against tumors, and it is not only necessary to activate the original immune system reaction in vivo, but also to maintain the duration and intensity of the reaction, which is the key to immunotherapy against tumors.The 2017 FDA approval of the immune checkpoint inhibitor PD-1 inhibitor pembrolizumab for patients with MSI-H / dMMR pan tumors laid the groundwork for immunotherapy in cholangiocarcinoma.In the current clinical study of advanced cholangiocarcinoma, the combination regimen of PD-1 inhibitor + FOLFOX4 / GEMOX demonstrated a favorable survival benefit with an acceptable safety profile in advanced cholangiocarcinoma.Tirelizumab (Baiji Shenzhou) is a humanized lgg4 anti programmed death receptor 1 (PD-1) monoclonal antibody designed to minimize binding to FC γ r receptors in macrophages.Preclinical data suggest that FC γ r receptor engagement in macrophages is followed by activation of antibody dependent cell-mediated killing of T cells, reducing the antitumor activity of PD-1 antibodies.Tirelizumab is currently under clinical investigation as a single agent and combination therapy worldwide, developing a range of broad indications for both solid tumours and haematological tumours.There are currently 15 potential registered clinical studies of bazea in China and worldwide, including 11 phase 3 studies, four pivotal phase 2 studies.A phase I / II study evaluating the efficacy of tirelizumab monotherapy in Chinese patients with advanced solid tumors across cancer types, using a 200 mg IV q3w dose and dosing schedule, has demonstrated tolerability at this dose in the Chinese population, a favorable clinical safety profile, and no contraindications in combination with chemotherapeutic agents such as capecitabine have been reported.

We plan to conduct a single center prospective interventional cohort study of capecitabine plus PD1 MAb given to patients who have been evaluated for high-risk recurrence after surgery for cholangiocarcinoma, to evaluate its efficacy and safety compared with capecitabine alone, and to strive for an effective treatment option in preventing postoperative metastatic recurrence of cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Post R0 resection, pathologically confirmed intrahepatic cholangiocarcinoma.Patients were also pathologically confirmed to have any of the following high-risk factors (ie, positive resection margins, positive lymph nodes, positive perineural invasion, and intrahepatic cholangiocarcinoma > 5cm in diameter;
* No history of any chemotherapy, radiotherapy, immunotherapy and interventional treatment prior to surgical resection;
* ECoG score 0-1 points;
* Liver function before medication child a, blood routine: WBC > 2.5 * 109 / L, PLT > 60 * 109 / L, coagulopathy: Pt prolonged < 2S, ALT < 150u / L;
* No heart, lung, or kidney function abnormalities were observed;
* No history of major bleeding disorders of the digestive tract;
* Signed informed consent;

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with other malignant tumor.
* Patients with mental illness.
* Patients participated in other clinical trials in last three months.
* Residual lesions showed by Postoperative digital subtraction angiography(DSA).
* Postoperative patients treated with other targeted drugs, PD1 antibody and other immunotherapies, FOLFOX systemic chemotherapy, and HuaiErKeLi drug treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
recurrence free survival (RFS) | 2 years
  the time from liver resection to tumor recurrence or metastasis

SECONDARY OUTCOMES:
Overall survival | 5 years
  the survival time after liver resection

CONTACTS AND LOCATIONS:
Locations (1):
- Lulu@Huashan.Org.Cn, Shanghai, China